CLINICAL TRIAL: NCT03031431
Title: Electricity-free Infant Warmer for Newborn Thermoregulation in Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Ministry of Health, Rwanda (Other Government); Rwandan Biomedical Counsel (RBC) (Unknown); Harvard Medical School (HMS and HSDM) (Other); Institute for Transformative Technologies (ITT) (Unknown); Brigham and Women's Hospital (Other); Partners in Health (Other)
Responsible Party: Principal Investigator, Anne Hansen, MD, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00016205
Record Dates: First submitted 2016-12-13; First posted 2017-01-25 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Hypothermia Neonatal
Keywords: Hypothermia; Infant Warmer
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Non-Electric Infant Warmer (Experimental): In line with current recommended practice, mothers will be encouraged to provide Kangaroo Mother Care (KMC) whenever possible. If an infant's temp is not rising by ½ degree C per hour with KMC alone, the infant warmer will be offered as an addition by the study team. If the mother is not available for KMC at any time, the infant will be warmed exclusively with the warmer. Bundling in clothes will only be used in addition to the warmer per carer preference. Temp measurement of the infant, warmer, and ambient air will be measured every 15 mins for the first hr, then hrly and as needed for the remainder of use or until warmer endpoint is reached (warmer temp below 36 degrees or phase-change material hardens [soft, semisoft, or hardened]).
  Interventions: Device: Non-Electric Infant Warmer

INTERVENTIONS:
Device: Non-Electric Infant Warmer — Electric warmers are the standard of care in developed countries, but are extremely costly, complicated with risk of causing both hypo and hyperthermia with misuse, and often not feasible in settings without stable electricity. Through a multi-institutional collaboration, the investigators have developed an electricity-free infant warmer.

SUMMARY:
Hypothermia contributes to a significant portion of neonatal deaths. Kangaroo mother care (KMC) is a safe and effective method of warming; however, it is not always feasible, and not possible in settings such as resuscitation or clinical instability. Electric warmers are the standard of care in developed countries, but are extremely costly, complicated with risk of causing both hypo and hyperthermia with misuse, and often not feasible in settings without stable electricity. Through a multi-institutional collaboration, the investigators have developed an electricity-free infant warmer. After laboratory based prototype testing for safety and efficacy, the investigators aim to study the supervised use of the warmer under routine implementation conditions in a resource-limited setting.

DETAILED DESCRIPTION:
Hypothermia contributes to a significant portion of neonatal deaths. Kangaroo mother care (KMC) is a safe and effective method of warming; however, it is not always feasible, and not possible in settings such as resuscitation or clinical instability. Electric warmers are the standard of care in developed countries, but are extremely costly, complicated with risk of causing both hypo and hyperthermia with misuse, and often not feasible in settings without stable electricity. Through a multi-institutional collaboration, the investigators have developed an electricity-free infant warmer. After laboratory based prototype testing for safety and efficacy, the investigators aim to study the supervised use of the warmer under routine implementation conditions in a resource-limited setting. The primary aim of Phase 1 is to determine if the infant warmer is a safe, effective, usable and functional addition to KMC. This is planned in a convenience sample of patients in two district hospitals, one in a relatively warm environment, and one in a colder setting using quantitative methods and observer audits of usability and functionality. After determination of safety and effectiveness and making any necessary modifications to the warmer, Phase 2 aims to study the warmer in rural health centers and transport, as this is where we ultimately aim to use the electricity free devices due to the limited access to functioning and stable electricity in these settings. The overall goal of the project is dissemination of the study results, and ultimately the infant warmer to the district and national level for key policy makers and stakeholders, as well as globally via publication.

ELIGIBILITY:
Inclusion Criteria:

* Any infant with the following criteria for whom caregiver is not available for Kangaroo Mother Care, or Kangaroo Mother Care is not adequate (less than ½ degree Celsius per hour rise in temperature).

  1. axillary temperature < 36 degrees C and ≥35 degrees C 1a) If an electric warmer is available and the infant's temperature is < 35 degrees C, then the infant would start by being warmed on the electric warmer until the infant's temperature reaches 36 degrees C, then can start non-electric infant warmer use
  2. Infants at-risk for hypothermia (criteria: estimated post-menstrual age of < 35 weeks or current body weight of < 2.5 kg)

Exclusion Criteria:

1. Any infant whose family is unwilling to consent to study.
2. Mothers who are critically ill at the time of infant eligibility or deemed not medically stable by nursing staff to be approached for consent.
3. Any infant with a contraindication to Kangaroo Mother Care (medical instability) and electrical heating source available.
4. Any infant with initial temperature < 35 degrees C and electrical heating source available.
5. Infants within the first hour of admission to neonatal unit or first hour of life in maternity.
6. Infants requiring phototherapy
7. Infants with significant skin condition
8. Infants with Hypoxic Ischemic Encephalopathy (HIE)

Stopping Criteria:

If an electric heating source is available, the infant will be taken off the study and warmed with an appropriate source of electric heat if the infant:

1. Is hypothermic and temperature decreases on any measurement
2. Is hypothermic and temperature does not begin to rise within 30 minutes
3. Is hypothermic and not heating at a rate of > ½ degree C per hour until temperature is >36.5 degrees C
4. Has a temperature that falls below 36 degrees C despite maximum exposure to the heat source
5. Is ever considered to be too severely ill by the medical team to be safely cared for in the non-electric infant warmer.
6. The warmer will be removed once its temperature drops below 36 degrees, and/or the phase change material begins to harden.

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2016-07; Primary Completion 2018-12 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Hansen, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Dr Evrard Nahimana, Rwinkwavu, Rwanda

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Encounters
Period: Overall Study
Arm/Group | Non-Electric Infant Warmer
Started | 130; 204 Encounters
Completed | 129; 203 Encounters
Not Completed | 1; 1 Encounters
Not completed — Infant removed by maternal request | 1

BASELINE CHARACTERISTICS:
Arm/Group | Non-Electric Infant Warmer
Number analyzed (Participants) | 130
Age, Customized [Count of Participants; unit: Participants]
  <37 weeks Gestation | 21
  >=37 weeks gestation | 51
  Missing/Not Known | 58
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Sex/Gender was not obtained or assessed
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Rwanda | 130
Birth Weight [Count of Participants; unit: Participants]
  ≥2500 g | 15
  1501 g to ≤2500 g | 96
  1001 g to ≤1500 g | 15
  ≤1000 g | 1
  Missing | 3
Age at First Encounter [Count of Participants; unit: Participants]
  1-7 days | 29
  8-31 days | 16
  32 days or more | 8
  On Birthday | 77

OUTCOME MEASURES:

1. Primary Outcome: Temperature/Effectiveness
Description: The infant warmer will be evaluated on the number of time is able to successfully achieve and maintain a normal body temperature for patients who are hypothermic and those patients at risk of hypothermia because of a < 2.5 kg birth weight or < 35 week gestational age.
Time Frame: Up to 6 months
Measure: Number; unit: Number of infant warmer uses
Units Other Than Participants: Encounters
Arm/Group | Non-Electric Infant Warmer
Number analyzed (Participants) | 130
Number analyzed (Encounters) | 204
Number of infant warmer uses
  Successfully reaches/maintains healthy temperature | 179
  Fails to reach/maintain healthy temperature | 4
  Not recorded | 21

2. Secondary Outcome: Usability
Description: The investigators will use observation to evaluate the usability of the warmer by assessing whether or not the infant warmer was used in a way that deviated from its recommended use.
Time Frame: Up to 6 months
Measure: Number; unit: Encounters with non-electric warmer
Units Other Than Participants: Encounters
Arm/Group | Non-Electric Infant Warmer
Number analyzed (Participants) | 130
Number analyzed (Encounters) | 204
Encounters with non-electric warmer
  Deviation from recommended use | 0
  No deviation from recommended use | 204

3. Secondary Outcome: Functionality
Description: The functionality will be assessed by whether or not there appeared to be wear and tear on the infant warmer based on repeated use.
Time Frame: Up to 6 months
Measure: Number; unit: infant warmers
Units Other Than Participants: Infant Warmers
Arm/Group | Non-Electric Infant Warmer
Number analyzed (Participants) | 103
Number analyzed (Infant Warmers) | 12
infant warmers
  Showed wear and tear | 5
  No wear and tear | 7

4. Secondary Outcome: Qualitative Survey
Description: The same as primary outcome and secondary outcome as described above with the setting being clinic and transport based rather than in a hospital, and with the addition of qualitative questions for mother and nurse regarding infant warmer use.
Time Frame: Up to 1 year
Population: Zero participants were analyzed as the investigators ultimately decided not collect qualitative data.
Arm/Group | Non-Electric Infant Warmer
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Non-Electric Infant Warmer
All-Cause Mortality (participants affected / at risk) | 0/130
Serious Adverse Events (participants affected / at risk) | 0/130
Other Adverse Events (participants affected / at risk) | 0/130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2015-02-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT03031431/Prot_ICF_000.pdf